CLINICAL TRIAL: NCT03348267
Title: Effect of Milk Protein Supplementation on Muscle Recovery and Football-specific Performance During an In-season Microcycle With Two Matches
Brief Title: Protein Supplementation and Muscle Recovery in Football
Acronym: PRO-FOOTBALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PROTEIN-FOOTBALL RECOVERY-UTH
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Skeletal Muscle Damage; Muscle Inflammation; Muscle Recovery; Soccer Performance
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein (Experimental): On the match day, 25g of protein consumed immediately after the match and then 30g at 3h (+3h) and 25g at 6h (+6h). On each day of the remaining days, 20 g of protein consumed with breakfast.
  Interventions: Dietary Supplement: Milk protein isolate
- Placebo (Active Comparator): On the match day, 500 ml received received orally immediately post-match and then at +3h and +6h. On the remaining days, 500 ml daily with breakfast.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Milk protein isolate — Milk protein isolate in a powder form consisted of 80% casein and 20% whey protein. 20g were diluted into 500 ml water
  Arms: Protein
Dietary Supplement: Placebo — 500 mL drink that contained water (375 mL), sugar-free cordial (125 mL) and 2 g of low-calorie glucose/dextrose powder.
  Arms: Placebo

SUMMARY:
Soccer is an intermittent sport including a high number of powerful actions such as accelerations, decelerations, changes of direction, jumps and impacts that incorporate a strong eccentric component and may therefore lead to skeletal muscle damage. Indeed, match activity is associated with the onset of muscle damage and an acute inflammatory response that result in attenuated performance for as long as 1 to 3 days. In competitive soccer though, multiple matches are performed within a small-time frame resulting in inadequate muscle recovery and reduced field performance. Supplementation with milk proteins following intense exercise protocols has been shown to stimulate protein synthesis and facilitate muscle recovery. Thus, the aim of the present investigation is to examine the effects of milk protein supplementation on muscle recovery and soccer-specific performance during an in-season microcycle with two matches performed three days apart.

DETAILED DESCRIPTION:
In a double-blind, cross over, repeated measures design 20 men soccer players will receive either placebo (PLA) or milk protein isolate (PRO, 80% casein-20% whey) throughout recovery following two matches performed three days apart. On match days, players will receive a dose immediately after the match (PLA vs PRO: 25g of protein) and then at 3h (PLA vs PRO: 30g of protein) and 6h (PLA vs PRO: 25g of protein) post-match. On each day of the remaining days, players will consume a single dose of PLA or PRO (20g of protein) with breakfast. All players will participate in regular in-season training following matches. Field activity during both matches and daily practices will be monitored using GPS devices. Heart rate will be continuously recorded during each match and training session. Blood samples will be collected at baseline as well as 2 hours after the first match, daily for three days after the first match, 2 hours after the second match and daily for 3 days after the second match. Performance (isokinetic strength, 20-m speed, repeated sprint ability) and muscle soreness will be assessed at baseline daily for 3 days after both matches. Muscle biopsies from vastus lateralis will be collected at baseline and one day after each match.

ELIGIBILITY:
Inclusion Criteria:

* i) participation at elite level (top three division leagues) of soccer competition for at least five years, ii) abstain from consumption of performance-enhancing supplements, antioxidant supplements and medications (for at least 6 months before and during the study), iv) participate in at least six two-hour training sessions per week and played at least one match per week and v) non-smokers.

Exclusion Criteria:

* i) a known milk intolerance or allergy, ii) a recent febrile illness, iii) history of muscle lesion, iv) lower limb trauma and v) metabolic diseases.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Change in creatine kinase in plasma | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Concentration of creatine kinase will be measured in plasma
Change in uric acid in plasma | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Concentration of uric acid will be measured in plasma
Change in protein carbonyls in blood | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Concentration of protein carbonyls will be measured in red blood cells
Change in total antioxidant capacity | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Total antioxidant capacity will be measured in plasma
Change in reduced glutathione in blood | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Concentration of reduced glutathione will be measured in in red blood cells
Change in oxidized glutathione in blood | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Concentration of oxidized glutathione will be measured in red blood cells
Change in malondialdehyde in blood | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Concentration of malondialdehyde will be measured in serum
Change in catalase activity | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Catalase activity will be measured in red blood cells
Change in protein carbonyls in muscle | At baseline, 24h post-Match 1 and 24h post-Match 2
  Concentration of protein carbonyls will be measured in muscle
Change in intracellular signaling proteins in muscle | At baseline, 24h post-Match 1 and 24h post-Match 2
  Phosphorylation levels of Akt, mammalian target of rapamycin (mTOR) and p70S6K will be measure using western blotting.
Change in proteasome activities in muscle | At baseline, 24h post-Match 1 and 24h post-Match 2
  Chymotrypsin-like (CT-L), caspase-like (C-L) and trypsin-like (T-L) proteasome activities will be assayed with hydrolysis of the fluorogenic peptide LLVY-AMC, LLE-AMC and LSTR-AMC, respectively.
Change in satellite cells in muscle | At baseline, 24h post-Match 1 and 24h post-Match 2
  Pax7, Myf5, MyoD and Myogenin will be measured in order to quantify quiescent, activated, proliferated-differentiated and fused satellite cells respectively.
Change in repeated Sprint Ability | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  5 x 30 m sprints will be performed with 25 seconds rest in-between. Mean time for 5 sprints and fatigue index will be calculated.
Change in countermovement jump | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Countermovement jump will be assessed on a contact platform
Change in isokinetic strength of lower limbs | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Isokinetic strength will be assessed on an isokinetic dynamometer for both knee extensors and knee flexors at 120 and 180 degrees.
Change in match activity | During Match 1 and Match 2
  Match activity will be continuously recorded during both matches using GPS technology.
Change in heart rate | During Match 1 and Match 2
  Heart rate will be continuously recorded during both matches using the Team Polar system.

SECONDARY OUTCOMES:
Change in delayed onset of muscle soreness | At baseline, at 24h, 48h and 72h post-Match 1 as well as at 24h, 48h and 72h post-Match 2
  Muscle soreness will assessed during palpation of the muscle belly and the distal region of relaxed vastus medialis, vastus lateralis and rectus femoris following three repetitions of of a full squat. Subjects will rate their DOMS on a visual analogue scale (0-10).
Dietary intake | Over a 7-day period at baseline.
  Dietary intake will be assessed using 7-day diet recalls.
Change in white blood cell count. | At baseline, immediately after Match 1, at 24h, 48h and 72h post-Match 1 as well as immediately after Match 2 and at 24h, 48h and 72h post-Match 2.
  White blood cell count will be measured using an automatic blood analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: ATHANASIOS POULIOS, PhDc, Principal Investigator — UNIVERSITY OF THESSALY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Trikala, Greece